CLINICAL TRIAL: NCT01827410
Title: High Agreement Between the Danish Ventral Hernia Database and Hospital Files in Region Zealand
Status: Completed | Type: Observational
Sponsor: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Frederik Helgstrand, MD, Zealand University Hospital
Other Study IDs: FH10
Record Dates: First submitted 2013-04-04; First posted 2013-04-09 (Estimated); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Data Agreement Between a Database and Hospital Files After a Ventral Hernia Repair

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients with a ventral hernia repair: All patients with a ventral hernia repair performed in Region Zealand and registered in The Danish Ventral Hernia Database during October 1st 2010 to October 1st 2011
  Interventions: Procedure: Ventral hernia repair

INTERVENTIONS:
Procedure: Ventral hernia repair

SUMMARY:
Is there agreement between data in the Danish Ventral Hernia Database and patient files

ELIGIBILITY:
Inclusion Criteria:

* All ventral hernia repairs

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hernia repairs performed in Region Zealand and registered in the Danish Ventral Hernia Database during the study period
Sampling Method: Non-Probability Sample
Enrollment: 408 (Actual)
Dates: Start 2010-10; Primary Completion 2011-10 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Data agreement | 1 year
  Compare information registered in The Danish Ventral Hernia Database with information obtained from patient files

CONTACTS AND LOCATIONS:
Overall Officials: Frederik Helgstrand, MD, Principal Investigator — Dept. Surgery, Køge Hospital, University of Copenhagen
Locations (1):
- Dept. of Surgery, Køge Hospital, Køge, Denmark